CLINICAL TRIAL: NCT05713565
Title: A Randomized-controlled Trial Evaluating a Digital Care Solution (Sidekick, SK-121) for Coronary Artery Disease Patients at Landspítali University Hospital
Brief Title: A Digital Care Solution for Coronary Artery Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidekick Health (Industry)
Collaborators: Landspitali University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SK-121-CAD
Record Dates: First submitted 2023-01-25; First posted 2023-02-06 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2023-02

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; digital application; lifestyle change; remote monitoring; clinical outcome; quality of life
MeSH Terms: conditions — Coronary Artery Disease | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Single center prospective randomized open blinded end-point (PROBE)
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded for group assignment at the 6-, and 12-month follow-up visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital Care Solution group (Experimental): Participants will be instructed to download the SKH mobile app to which the participants will have access for 12 months, and the participants will receive an access code to activate the SKH CAD program. The aim of the program is to empower self-assessment of CAD symptoms as well as positive lifestyle change by gamification, altruistic rewards, and engaging content with relevant tasks or missions to be completed.
  Beyond this, all patients in the interventional arm will also receive standard of care as defined below for the control arm.
  Interventions: Device: A digital care solution for patients with Coronary Artery Disease; Other: Standard of care for patients with Coronary Artery Disease
- Standard of Care - control group (Active Comparator): The participants in the Standard of Care - control group will receive an information leaflet about relevant lifestyle modifications for CAD. After baseline measurements and data collection, follow-up and continuous care will be as usual in outpatient care (i.e., Standard of Care).
  Interventions: Other: Standard of care for patients with Coronary Artery Disease

INTERVENTIONS:
Device: A digital care solution for patients with Coronary Artery Disease — A digital care solution that provides remote patient monitoring and a patient support program specifically developed for CAD patients. The digital care solution empowers self-assessment of CAD symptoms as well as positive lifestyle change by gamification, altruistic rewards, and engaging content with relevant tasks or missions to be completed.
  Other Names: SK-121
  Arms: Digital Care Solution group
Other: Standard of care for patients with Coronary Artery Disease — Follow-up and continuous care as usual in outpatient care (i.e., Standard of Care). The participants in the Standard of Care - control group will also receive an information leaflet about relevant lifestyle modifications for CAD.

SUMMARY:
This is a single center, randomized clinical trial (RCT), recruiting 200 patients with coronary artery disease (CAD) who are currently receiving standard care treatment at the cardiology department of Landspítali University Hospital in Reykjavik, Iceland.

The RCT will determine whether an interactive health app that supports lifestyle changes can positively impact disease progression and quality of life of CAD patients. Patients will be randomized to receive either the standard of care (SoC) alone or SoC with the addition of the digital app. The digital app will include remote patient monitoring and a patient support program specific for CAD patients.

The investigators will study the impact of the digitally delivered lifestyle intervention and remote monitoring on disease progression and on the patients' quality of life.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of death worldwide, with an estimated number of 17.9 million deaths each year. Coronary artery disease (CAD) is the most common form of CVD and is caused by plaque buildup (atherosclerosis) in the walls of the coronary arteries that supply blood to the heart. The plaques consist of deposits of cholesterol, fat, calcium and other substances. Atherosclerosis of the coronary arteries reduces blood flow to the heart and can eventually result in a myocardial infarction.

Lifestyle-related risk factors are known to play an important role in the development of CAD and CVD in general and many of these risk factors are modifiable. The most important modifiable cardiovascular risk factors are an unhealthy diet, physical inactivity, smoking use, and excessive use of alcohol. Improvements in these modifiable risk factors can significantly lower the risk of recurrent events in CVD patients.

Many clinical trials have shown that lifestyle interventions focused on for instance improving diet, physical activity, weight and waist circumference reduce cardiovascular risk scores. Also, recurrence of cardiac events can be reduced by lifestyle interventions as smoking cessation was associated with 43% reduction of recurrent myocardial infarction, and regular exercise and diet modifications reduced the risk of recurrent myocardial infarction by 48%. Exercise intervention reduced mortality by 27% and diet intervention reduced mortality by 26%. While on the other hand reduced physical activity has been shown to increase the risk of cardiac death in CAD patients.

Lifestyle modification has not only been shown to improve quality of life but is also cost-effective. Lifestyle intervention is recommended by clinical guidelines, but a gap exists between recommendations and what is being implemented in clinical practice. Finding simple ways to incorporate lifestyle intervention to standard CAD care could undoubtedly improve patient outcomes and the disease burden.

Because of the widespread ownership of smartphones, digital applications hold promise for providing lifestyle modification support to large numbers of people in a format that is readily accessible at almost any time. Approximately two-thirds of the world's population owns a smartphone, and in 2019 there were 204 billion app downloads. Considering the evidence, the use of digital applications seems supported. However, currently, there is still limited data to draw from on the effectiveness of digitally delivered remote monitoring and patient support programs for CAD patients. As a result, more data is needed.

In this study, Sidekick Health's newly developed digital care solution, including remote patient monitoring (RPM) and a patient support program (PSP) specifically developed for CAD patients, will be tested. Comparing the effect of adding a digital solution to the standard of care (SoC), this study will investigate the impact of a holistic, digitally delivered lifestyle intervention and remote monitoring on disease progression and on the CAD patient's quality of life.

The aim of this study is to test the effectiveness of improving clinical outcomes and quality of life by using the Sidekick Health's CAD digital program in combination with SoC compared to SoC alone.

ELIGIBILITY:
Inclusion Criteria:

* Adults diagnosed with coronary artery disease
* Fluent in verbal and written Icelandic
* Capacity to give informed consent
* Capacity to operate a smartphone

Exclusion Criteria:

* Not owning a smartphone compatible with the Sidekick Health app or not willing to have it installed on their device
* Not able or willing to comply with study intervention/scheduled measures and visits
* Having another serious medical condition (e.g., cancer, endocarditis, heart failure (EF<40%), history of cardiac arrest)
* Active alcohol or drug abusers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Risk of recurrent Coronary Artery Disease | 12 months
  Difference in change in total score of the Second Manifestations of ARTerial disease (SMART) risk score between the intervention and control groups.
  The SMART Risk Score is based on 13 demographic and clinical parameters, the resulting SMART Risk Scores range from 0 to 100%, with a lower score representing a lower risk.

SECONDARY OUTCOMES:
CAD-specific health status | 12 months
  Difference in change in the total score of the 7-item Seattle Angina Questionnaire - 7 (SAQ-7) between the intervention and control groups.
  The SAQ-7 consists of a self-reported list with 7 questions (1a-c and 2-5) where one can choose between six (questions 1a to 3) or five (questions 4 and 5) answers by ticking boxes. The answers of 1a and 1b are on Likert scales where 1 represents "extremely limited" to 6 "limited for other reasons or did not do the activity". The answers of 2 and 3 are on Likert scales where 1 represents "4 or more times per day" to 6 "none over the past 4 weeks". The answers of question 4 are on a Likert scale where 1 represents "it has extremely limited my enjoyment of life" to 5 "it has not limited my enjoyment of life at all". The answers of question 5 are on a Likert scale where 1 represents "not satisfied at all" to 5 "completely satisfied". Scores are on a scale of 7 to 39 with low scores denoting the worst and high scores the best possible status.
Burden of Coronary Artery Disease | 12 months
  Difference in burden of Coronary Artery Disease between intervention and control group as measured by (costs of) number of Coronary Artery Disease-related visits to emergency room, hospital, and the cardiology department.
Medication adherence | 12 months
  Difference in self-assessed medication adherence between intervention and control group as measured by the 8-item Morisky Medication Adherence Scale (MMAS-8).
  The MMAS-8 is an 8-item structured, self-reported medication adherence measure. The total score on the MMAS-8 has a range from 0 to 8.0. The 3 categorical Likert Scale is: low adherence is <6, medium adherence is 6 to <8, and high adherence is 8.
Patients self-care and disease knowledge | 12 months
  Difference in self-care and disease knowledge between intervention and control group as measured by the self-assessed Coronary Artery Disease Education Questionnaire - Short Version (CADE-Q SV).
  The CADE-Q SV is a 20-item questionnaire where one can choose between three answers by ticking boxes "True", "False", or "I don't know". Each correct answer is given 1 point. The scores on the CADE-Q SV range from 0 to 20, with low scores denoting the worst and high scores the best possible self-care and disease knowledge.
Smoking status | 12 months
  Difference between intervention and control group in self-reported smoking status
Depression, anxiety, and stress levels | 12 months
  Difference in change in the total score of the 21-item Depression, Anxiety and Stress Scale (DASS21) questionnaire between the intervention and control group.
  Each question on the DASS21 has a Likert scale of 4 options where 0 represents "did not apply to me" to 3 "applied to me very much". The scores on the subscales range from 0 to 63, and low scores indicate a better mental health status.

CONTACTS AND LOCATIONS:
Overall Officials: David O Arnar, MD, PhD, Principal Investigator — National University Hospital of Iceland & University of Iceland
Locations (1):
- Landspítali University Hospital, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: No
Anonymized Individual Participant Data may be shared with other researchers for relevant research purposes following complementary ethical review and approval from the Ethical Review Board.